CLINICAL TRIAL: NCT01923766
Title: Adoptive Transfer of Cord Blood T Cells to Prevent and Treat CMV, EBV and Adenovirus Infections After Transplantation
Brief Title: Cytotoxic T Cells to Prevent Virus Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Catherine Bollard, Director- Center for Emerging Technologies in Immune Cell Therapies (CETI), Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTCAT2
Record Dates: First submitted 2013-08-08; First posted 2013-08-16 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: CMV; EBV; Adenovirus Infections
Keywords: Transplantation
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cytotoxic T lymphocytes (CTLs) (Experimental): Cytotoxic T lymphocytes (CTLs). CMV/AdV /EBV specific T cells will be given by slow intravenous injection over 1-2 minutes. Four dose levels will be explored. The lowest dose level will be 5x106cells/m2 and the highest will be 2.5x107/m2. During the dose escalation phase two to six patients will be entered at each dose level (depending on toxicity). If there are no toxicities and immunological efficacy is not seen at any dose, then the doses will be further escalated after additional local and federal approval.
  Interventions: Drug: Cytotoxic T lymphocytes (CTLs).

INTERVENTIONS:
Drug: Cytotoxic T lymphocytes (CTLs). — This Phase I dose-escalation trial is designed to evaluate the safety of donor-derived cytotoxic T lymphocytes (CTLs). Dose escalation is guided by the modified continual reassessment method (mCRM) in order to determine the maximum tolerated dose (MTD). For each group, MTD is defined as the dose at which the probability of DLT is at most 21%. Four dose levels are being evaluated namely, 5x106 cells/m2, 1.0x107 cells/m2, 1.5x107 cells/m2 and 2.5x107 cells/m2 with prior probabilities of toxicity estimated at 5%, 7.1%, 10% and 21%, respectively.
  Two patients are allocated in each cohort and are followed for 30 days post IV injection for evaluation of DLTs. The trial continues until a minimum of 12 patients have been treated and stop when the maximum 18 patients have been treated.

SUMMARY:
In this study, investigators are trying to see if infusion of "m-CTLs" will prevent or treat cytomegalovirus (CMV), Epstein Barr Virus (EBV) and adenovirus (AdV) reactivation or infection after cord blood transplant.

Patients with blood cell cancer, other blood disease or a genetic disease may receive a cord blood transplant (UCBT) from an unrelated donor. After receiving a cord blood transplant, they are at risk of infections until a new immune system to fight infections grows from the cord blood cells. In this study, investigators are trying to give special cells from the cord blood called T cells. These cells will try to fight viruses that can cause infection.

Investigators will test to see if blood cells from donor that have been grown in a special way, can prevent patients from getting an infection. EBV, AdV and CMV are viruses that can cause serious life-threatening infections in patients who have weak immune systems after transplant.

T lymphocytes can kill viral cells but normally there are not enough of them to kill all the virus infected cells after transplant. Some researcher have taken T cells from a person's blood, grown more of them in the laboratory and then given them back to the person during a viral infection after a bone marrow transplant. Some of these studies have shown a positive therapeutic effect in patients receiving the CTLs (specially trained T cells) after a viral infection in the post-transplant period. In this study we are trying to prevent or treat viral infections by given the CTLs soon after getting the umbilical cord blood transplant.

With this study, investigators want to see if they can use a kind of white blood cell called T cells to prevent or treat AdV, EBV and CMV infection. Investigators will grow these T cells from the cord blood before transplant. These cells have been trained to attack adenovirus/EBV/CMV- infected cells and are called multivirus-specific cytotoxic (killer) T-cells or "m-CTL." Investigators would plan to give patients one dose of m-CTL any time from 30 to 364 days after your transplant. They have used T cells made in this way from the blood of donors to prevent infections in patients who are getting a bone marrow or blood stem cell transplant but this will be the first time investigators make them from cord blood.

DETAILED DESCRIPTION:
Umbilical cord blood (UCB) is a readily available alternative source of Hemotopoietic Stem Cells (HSCs) that is capable of reconstituting hematopoiesis after myeloablative therapy. More than 280,000 UCB units have been banked world-wide and more than 13,000 unrelated donor UCB transplantations have been performed.

UCB transplants offer several advantages over adult bone marrow or peripheral blood stem cell transplants, including: 1) rapid availability, 2) absence of donor risk, 3) low risk of transmissible infectious diseases, 4) low risk of acute Graft versus Host Disease (GvHD) in the setting of Human Leukocye Antigen (HLA) mismatch (as compared to recipients of unrelated donor marrow and peripheral blood). UCB is particularly beneficial for patients of ethnic and racial minority descent for whom adult marrow and blood donors often cannot be identified.

In a larger series the neutrophil engraftment has been reported as high as 92%. The incidence of acute GvHD reported in larger series ranges from 33-44% to 11-22% for grades II-IV and III-IV acute GvHD, respectively. The incidence of chronic GvHD ranges from 0-25%. These results are particularly notable since most UCB donor-recipient pairs are 1-2 HLA antigen mismatched. However, infection related TRMs are still of concern after UCBT. The rate of hemopoietic recovery is slower after UCBT; therefore infectious complications including viral infections occur frequently.

Multi virus Specific T cells from Cord Blood could be applied with comparable success to recipients of CB transplants; however, certain obstacles to the extension of this approach must be circumvented. These include: (i) the limited numbers of CB T-cells available for manipulation and (ii) the naivety of CB T-cells. Hence, the development of virus-protective T-cell therapy for patients undergoing CBT requires the priming and extensive expansion of naïve T-cells rather than the more limited and simple direct expansion of pre-existing virus-specific memory T-cell populations from virus-experienced donors. Further, CB T-cells have lower cytotoxic activity and higher activation-induced cell death than peripheral blood T-cells. These limitations have prevented the production of virus-specific cord blood-derived CTL in sufficient numbers for clinical use. Because of these challenges, only a few reports document the generation of antigen-specific T cells from CB. Sun et al first reported the ability to generate EBV-specific CD4+ T cells using EBV-transformed B-cells, or lymphoblastoid cell lines (LCL). Park et al then reported the ability to generate CMV-pp65-specific T cells from cord blood by using CMV-immune complex-loaded DCs, CMV lysate, and IL-12 and IL-7. The study at Baylor College of Medicine (BCM)showed that Ad5f35pp65-transduced CB-derived APC could be used to generate large numbers of autologous T-cells specific for both CMV and Ad, even from the phenotypically naive T-cell subpopulation. Addition of EBV-transformed B-lymphoblastoid cell lines (LCL) to the APCs allowed the Ad/CMV specificity of the CB T-cells to be extended to EBV. In addition, the multivirus-specific T-cells recognized an array of epitopes after only 2 weeks expansion in vivo. We therefore suggest that our ability to generate virus-specific CTL from CB against a plethora of epitopes recognized by both CD4+ and CD8+ T-cells should minimize the risk of viral escape and maximize therapeutic benefit on administration of these cells to cord blood recipients at risk of severe viral disease. A clinical trial using CB-derived multi-virus specific T cells for the prevention and treatment of viral infection after CBT was started at BCM. (Clinical Trial #: NCT01017705).

ELIGIBILITY:
Inclusion criteria at the time of Procurement:

* Patient with malignant or nonmalignant diseases who are candidates for transplant.
* Patients must have a CB unit (or units) matched with the patient at 4, 5, or 6/6 HLA class I (serological) and II (molecular) antigens.

Inclusion criteria at the time of CTL infusion:

* Recipients of at least one unmanipulated cord blood unit fractionated into 2 fractions (i.e. from a HLA matched or mismatched unrelated donor) transplant at risk for or with CMV/Adenoviral disease or reactivation.
* Lansky/Karnofsky scores >60
* Absolute neutrophil count (ANC) greater than 500/ul.
* No evidence of GVHD > Grade II at time of enrollment.
* Life expectancy > 30 days
* Absence of severe renal disease (Creatinine > x 3 normal for age)
* Absence of severe hepatic disease. Direct bilirubin must be < 3 mg/dl and AST < 5x upper limit of normal.
* Patient must be at least 30 days post transplant to be eligible to receive CTL
* Written informed consent and/or signed assent line from patient, parent or guardian.
* Patient not on Fi02 of >60%

Exclusion criteria at the time of Procurement

* Pregnant or lactating
* Patients with active central nervous system disease
* Patients with Karnofsky performance status <70%
* Patients with grade 3 or 4 or primary myelofibrosis
* Patients with suitable related donors

Exclusion criteria at the time of CTL infusion

* Pregnant or lactating
* Unable to wean steroids to ≤0.5 mg/kg/day prednisone.
* Patients with other uncontrolled infections (except CMV and/or adenovirus and/or EBVemia).
* Patients with less than 50% donor chimerism in either peripheral blood or bone marrow or patients with relapse of original disease.

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
To assess the safety of administration of CTLs | At 45 days post-infusion
  The primary endpoint is to assess the safety of administration of CTLs at 45 days post-infusion. The safety endpoint will be defined as acute GvHD grades III-IV or grade 3 or higher toxicity. Other toxicities to consider include GI , renal , hemorrhagic , cardiovascular, neurologic toxicity, coagulation, vascular and pulmonary toxicity.
  For the trial, two patients are allocated in each cohort and are followed for 45 days post IV injection of virus-specific T-cells for evaluation of DLTs. A maximum 18 patients will be accrued into each group. The final maximum tolerated dose (MTD) will be the dose with probability closest to the target toxicity rate at these termination points. The trial continues until a minimum of 12 patients have been treated. The trial will stop when the maximum 18 patients have been treated, or when six patients have been treated at the current MTD. We therefore expect to enroll between 12-18 patients into this trial.

SECONDARY OUTCOMES:
Viral load | Viral load will be monitored before infusion and after infusion weekly for a total of 60 days.
  Viral load will be monitored using PCR amplification. AdV surveillance cultures, or PCR studies in patients with positive AdV pre CTL will be taken before infusion and then weekly for 60 days.
  Patients will be monitored using ELISPOT assays or tetramer assays with appropriate viral specific peptide mixtures if sufficient cell numbers and appropriate reagents are available.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Bollard, M.D, Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Amanda Olson, MD, Houston, Texas